CLINICAL TRIAL: NCT01677377
Title: A Phase 2A, Open-Label, Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Primary Pharmacodynamic Markers of Efficacy of 60mg, 90mg, and 120mg of Risperidone in RBP-7000 Subcutaneous Injections in Subjects With Clinically Stable Schizophrenia
Brief Title: Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetic/Efficacy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-09-0009
Record Dates: First submitted 2012-08-27; First posted 2012-09-03 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic; Schizophrenias
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1, RBP-7000 60 mg (Experimental): Participants who were stable on 2 mg oral daily risperidone during the run-in period received 3 single,unblinded, subcutaneous (SC) injection doses of 60 mg risperidone in RBP-7000 on study days 1, 29 and 57. Participants returned to 2 mg oral daily risperidone on days 85-87.
  Interventions: Drug: Risperidone; Drug: RBP-7000
- Cohort 2, RBP-7000 90 mg (Experimental): Participants who were stable on 3 mg oral daily risperidone during the run-in period received 3 single,unblinded, subcutaneous (SC) injection doses of 90 mg risperidone in RBP-7000 on study days 1, 29 and 57. Participants returned to 3 mg oral daily risperidone on days 85-87.
  Interventions: Drug: Risperidone; Drug: RBP-7000
- Cohort 3, RBP-7000 120 mg (Experimental): Participants who were stable on 4 mg oral daily risperidone during the run-in period received 3 single,unblinded, subcutaneous (SC) injection doses of 120 mg risperidone in RBP-7000 on study days 1, 29 and 57. Participants returned to 4 mg oral daily risperidone on days 85-87.
  Interventions: Drug: Risperidone; Drug: RBP-7000

INTERVENTIONS:
Drug: Risperidone — Oral risperidone was supplied as 2, 3, or 4 mg tablets in blister packs or bottles and taken daily only during the oral dosing periods of the study, days -14 through -8 (if applicable), days -7 through -1, and days 85 through 87.
  Other Names: Risperdal
Drug: RBP-7000 — RBP-7000 60 mg, 90 mg, and 120 mg were a mixture of the ATRIGEL® Delivery System and 60 mg, 90 mg, or 120 mg risperidone, respectively. Treatment was delivered as subcutaneous injections on study days 1, 29 and 57.
  Other Names: risperidone in Atrigel

SUMMARY:
Evaluate the safety and tolerability of multiple subcutaneous injections of various dosages of risperidone with clinically stable schizophrenia

DETAILED DESCRIPTION:
This will be an open-label, Phase 2A, multiple ascending dose study in 1 to 3 sites, designed to evaluate the safety, tolerability, and pharmacokinetic (PK) profile of multiple subcutaneous injections of 60mg, 90mg, and 120mg doses of risperidone in the RBP-7000 formulation, in subjects with clinically-stable schizophrenia who are on a once daily stable dose of 2mg, 3mg, or 4mg of oral risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* > 18 to < 65 years
* Diagnosis of paranoid, residual, or undifferentiated schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR) criteria

  * Status: clinically stable subjects defined as subjects with no hospitalizations for acute exacerbations within 3 months of screening and screening total Positive and Negative Syndrome Scale (PANSS) score < 60
* Subjects who have given written informed consent

Exclusion Criteria:

* Subjects taking any risperidone sustained release formulation within the 60 days prior to study screening
* Subjects taking the following concurrent medication/over-the-counter products:
* Inducers or inhibitors of cytochrome P450 2D6 (CYP-2D6) within 14 days or 7 half - lives (whichever occurs last) prior to study screening
* Bupropion, chlorpheniramine, cimetidine, clomipramine, doxepin, or quinidine within 30 days prior to study screening
* Clozapine, phenothiazines, aripiprazole, haloperidol, or any other antipsychotic other than oral risperidone within 14 days prior to study screening
* Selective serotonin reuptake inhibitors (e.g., fluoxetine, paroxetine) or serotonin-norepinephrine reuptake inhibitors (e.g., venlafaxine, desvenlafaxine, duloxetine) within 30 days prior to study screening
* Opioids or opioid-containing analgesics within 14 days prior to study screening
* Medications, in addition to those listed above, which may be expected to significantly interfere with the metabolism or excretion of risperidone and/or 9-hydroxyrisperidone, that may be associated with a significant drug interaction with risperidone, or that may pose a significant risk to subjects' participation in the study
* Subjects with a history of cancer (with the exception of resected basal cell or squamous cell carcinoma of the skin) unless they have been disease free for >5 years
* Subjects with another active medical condition or organ disease that may either compromise subject safety and/or outcome evaluation of the study drug
* Subjects with evidence or history of a significant hepatic disorder that may either compromise subject safety or interfere with the safety and/or outcome evaluation of the study drug. Individuals with acute hepatitis (including but not limited to B or C); or individuals with 1) total bilirubin >1.5x the upper limit of normal and/or 2) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x upper limit of normal (ULN) will be excluded
* Subjects with hepatitis C antibody and AST, ALT, or alkaline phosphatase >2x and total bilirubin >1.3 mg/dL will be excluded
* Subjects with a history of renal disease, or a creatinine clearance of less than 80 mL/min (as determined by the Cockcroft Gault formula)
* Subjects with an international normalized ratio >2.0 at screening
* Subjects with corrected QT interval (Bazett's - QTcB) >450 msec (male) or >470 msec (female) at screening. Subjects with a QTc above these levels due to a benign right bundle branch block can be included in the study at the discretion of the PI
* Subjects who are known to have AIDS or to be HIV positive
* Subjects with suicidal ideation with intent and plan (Columbia-Suicide Severity Rating Scale (C-SSRS) affirmative answers to questions 4 and 5 of the ideation section) or suicide attempts within the last six months as noted on the C-SSRS, or subjects with uncontrolled depression in the opinion of the investigator
* Subjects with known diagnosis of type 1 or 2 diabetes or subjects with Hemoglobin A1c >7.0 at screening
* Subjects who have participated in a clinical trial within 30 days prior to study screening
* Subjects who meet the DSM-IV-TR criteria for alcohol abuse or dependence within the last six months of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Whitelaw, Sr. Dir of Proj Deliver, Study Director — Pharmaceutical Research Associates; Ashley Huston, PMP, Study Director — Pharmaceutical Research Associates
Locations (2):
- United States (2):
  - Woodland International Research Group, Inc., Little Rock, Alaska
  - Ocean View Psychiatric Health Facility, Long Beach, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, Phase 2A, multiple-ascending dose study performed at 2 sites in the U.S. Seventy subjects were screened and 45 subjects were enrolled and received RBP-7000.
Period: Overall Study
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Started | 15 | 15 | 15
Completed | 14 | 14 | 9
Not Completed | 1 | 1 | 6
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (9.98) | 42.5 (9.93) | 41.7 (7.96) | 42.6 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 1 | 12
  Male | 8 | 11 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 14 | 13 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 4 | 4 | 15
  Black or African American | 7 | 11 | 10 | 28
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 83.76 (16.279) | 84.07 (13.707) | 92.63 (14.075) | 86.82 (14.980)
Height [Mean (Standard Deviation); unit: cm] | 172.19 (8.731) | 175.50 (11.137) | 174.41 (8.346) | 174.03 (9.372)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.13 (4.487) | 27.35 (4.176) | 30.43 (3.911) | 28.64 (4.309)
Cytochrome P450 2D6 (CYP-2D6) [Count of Participants; unit: Participants] — CYP-2D6 is an enzyme responsible for the metabolism and elimination of many drugs. Considerable variation exists in the efficiency and amount of CYP-2D6 enzyme produced between individuals. Hence, for drugs that are metabolized by CYP-2D6, certain individuals will eliminate these drugs quickly (ultrarapid metabolizers) while others slowly (poor metabolizers).
  * poor metabolizer - little or no CYP-2D6 function
  * intermediate metabolizers - metabolize drugs at a rate somewhere between the poor and extensive metabolizers
  * extensive metabolizer - normal CYP-2D6 function
  Participants
    Intermediate | 3 | 0 | 1 | 4
    Poor | 1 | 1 | 0 | 2
    Extensive | 11 | 14 | 14 | 39

OUTCOME MEASURES:

1. Primary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any study-related event that represents a change (positive or negative) in frequency or severity from a baseline (prestudy) event (if any), regardless of the presence of causal relationship or medical significance. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the first study dose date. AEs are determined by the Investigator to be related or not related to the study drug.
  A serious AE (SAE) is defined by federal regulation as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Although a subject may have had 2 or more adverse experiences the subject is counted only once in a category. The same subject may appear in different categories.
Time Frame: Day 1 to Day 106
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
Participants
  No TEAEs | 4 | 4 | 7
  1 or more TEAEs | 11 | 11 | 8
  Related TEAEs | 6 | 11 | 4
  Serious TEAEs | 0 | 0 | 1
  Serious, related TEAE | 0 | 0 | 0
  TEAE causing discontinuation | 0 | 0 | 0
  Death | 0 | 0 | 0

2. Primary Outcome: Total Risperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24)
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  AUC0-24 calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: The PK analysis population was defined as all participants who received an injection of RBP-7000 and had an adequate number of PK blood draws (as determined by a clinical pharmacologist/pharmacokineticist) in order to provide a meaningful analysis of PK parameters.
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Initial Peak, Injection 1: number analyzed (Participants) | 14 | 15 | 15
  Initial Peak, Injection 1 | 335.4 [178.4 to 874.4] | 437.5 [203.2 to 942.3] | 466.2 [193.6 to 872.0]
  Initial Peak, Injection 3: number analyzed (Participants) | 13 | 12 | 8
  Initial Peak, Injection 3 | 276.5 [113.3 to 821.6] | 415.1 [151.4 to 697.0] | 497.5 [304.9 to 788.2]

3. Primary Outcome: Total Risperidone PK: Maximum Plasma Concentration (Cmax) During Initial Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Cmax determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Initial Peak, Injection 1 | 16.343 [8.49 to 45.33] | 19.415 [9.88 to 41.14] | 24.400 [9.00 to 42.71]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 14.549 [5.71 to 37.66] | 16.973 [7.06 to 39.44] | 22.852 [13.35 to 39.17]

4. Primary Outcome: Total Risperidone PK: Time of Maximum Plasma Concentration (Tmax) During Initial Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Tmax determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Initial Peak, Injection 1 | 6.000 [3.00 to 23.83] | 6.000 [2.00 to 12.02] | 6.000 [2.00 to 24.00]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 17.917 [6.00 to 24.00] | 24.000 [3.00 to 24.08] | 24.000 [6.00 to 24.00]

5. Primary Outcome: Total Risperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to Time Tau (Where Tau=28 Days) (AUCtau)
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  AUCtau calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 6506.0 [2400.2 to 16817.9] | 8293.8 [3680.3 to 19454.6] | 12594.7 [7894.8 to 17498.4]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 8567.1 [3890.3 to 17097.5] | 11047.7 [7197.5 to 22067.1] | 15982.6 [10256.6 to 18661.0]

6. Primary Outcome: Total Risperidone PK: Average Plasma Concentration (Cavg) Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The average of plasma concentrations calculated as AUCtau/ tau (tau = 28 days)
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 9.682 [3.57 to 25.03] | 12.342 [5.48 to 28.95] | 18.742 [11.75 to 26.04]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 12.749 [5.79 to 25.44] | 16.440 [10.71 to 32.84] | 23.784 [15.26 to 27.77]

7. Primary Outcome: Total Risperidone PK: Maximum Plasma Concentration (Cmax) Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Maximum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 16.878 [9.35 to 57.61] | 22.825 [10.89 to 41.14] | 32.235 [19.53 to 55.89]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 17.885 [8.56 to 42.11] | 30.804 [16.64 to 55.63] | 38.300 [23.76 to 53.45]

8. Primary Outcome: Total Risperidone PK: Minimum Plasma Concentration (Cmin) Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Minimum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 4.867 [1.88 to 13.54] | 5.642 [2.63 to 20.31] | 9.159 [3.28 to 15.23]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 5.028 [1.79 to 11.64] | 10.534 [3.85 to 14.80] | 11.938 [6.56 to 14.20]

9. Primary Outcome: Total Risperidone PK: Percent Fluctuation Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The degree of fluctuation of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cavg, expressed as a percentage.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 151.211 [69.88 to 371.07] | 135.238 [71.94 to 217.01] | 153.386 [64.60 to 179.59]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 108.226 [59.48 to 185.63] | 102.396 [57.34 to 162.19] | 114.008 [86.28 to 181.92]

10. Primary Outcome: Total Risperidone PK: Swing Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The swing of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cmin.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Overall, Injection 1 | 2.502 [1.02 to 12.44] | 2.150 [1.03 to 5.39] | 2.928 [0.98 to 8.40]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 2.588 [0.90 to 7.48] | 2.052 [0.74 to 4.29] | 2.019 [1.47 to 6.07]

11. Primary Outcome: Total Risperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the PK Profile
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Overall, Injection 1 | 168.000 [4.00 to 504.00] | 215.833 [4.00 to 579.02] | 192.000 [6.00 to 574.30]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 216.00 [12.00 to 408.00] | 264.067 [24.00 to 408.00] | 216.000 [168.00 to 504.18]

12. Primary Outcome: Total Risperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Area Under the Plasma Concentration Curve (Rac(AUC))
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Accumulation index in terms of AUC calculated as ratio of AUCtau injection 3 / injection 1. Tau = 28 days.
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 14 | 10
ratio | 1.1 [0.8 to 2.9] | 1.6 [1.0 to 2.9] | 1.2 [1.0 to 1.7]

13. Primary Outcome: Total Risperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Maximum Plasma Concentrations (Rac(Cmax))
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Accumulation index in terms of Cmax calculated as ratio of Cmax injection 3 / injection 1.
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 15 | 10
ratio | 0.976 [0.62 to 2.21] | 1.525 [0.73 to 2.83] | 1.105 [0.81 to 2.19]

14. Primary Outcome: Total Risperidone PK: Area Under the Plasma Concentration-Time Curve From Day 2-29 Post Injection (AUC Day 2-29)
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Area under plasma concentration-time curve from 24 hours (Day 2) to the last quantifiable collection during dosing interval (28 days); calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 at time of study drug administration.
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 6186.9 [2219.4 to 16241.8] | 7735.1 [3458.0 to 18517.4] | 10001.4 [5973.7 to 16936.7]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 8236.4 [3726.5 to 16278.8] | 10988.6 [7047.1 to 21379.3] | 15484.3 [9954.0 to 17931.7]

15. Primary Outcome: Total Risperidone PK: Average Plasma Concentration Over the Secondary Peak (Cavg, Day 2-29)
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The average of plasma concentrations in the plateau, calculated as AUC Day 2-29/time
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 9.548 [3.42 to 25.06] | 11.937 [5.34 to 28.58] | 15.434 [9.22 to 26.14]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 12.710 [5.75 to 25.12] | 16.958 [10.88 to 32.99] | 23.896 [15.36 to 27.67]

16. Primary Outcome: Total Risperidone PK: Maximum Plasma Concentration Over the Secondary Peak (Cmax)
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Maximum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  Secondary Peak, Injection 1 (Day 2 - Day 29) Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 16.867 [6.42 to 57.61] | 21.415 [9.26 to 41.06] | 32.235 [19.53 to 55.89]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 17.885 [8.56 to 42.11] | 30.804 [16.64 to 55.63] | 38.300 [23.76 to 53.45]

17. Primary Outcome: Total Risperidone PK: Minimum Plasma Concentration (Cmin) Over the Secondary Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Minimum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 4.867 [1.88 to 13.54] | 5.642 [2.63 to 20.31] | 9.159 [3.28 to 15.23]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 5.028 [1.79 to 13.33] | 10.534 [3.85 to 18.26] | 13.735 [8.47 to 21.91]

18. Primary Outcome: Total Risperidone PK: Percent Fluctuation Over the Secondary Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The degree of fluctuation of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cavg, expressed as a percentage.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 122.350 [70.17 to 246.65] | 122.042 [72.60 to 204.59] | 151.294 [76.81 to 187.04]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 101.788 [59.50 to 183.28] | 101.666 [55.92 to 162.53] | 96.489 [80.33 to 162.36]

19. Primary Outcome: Total Risperidone PK: Swing Over the Secondary Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  The swing of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cmin.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Secondary Peak, Injection 1 | 2.048 [1.02 to 12.44] | 2.017 [1.02 to 5.39] | 2.928 [0.98 to 5.26]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 2.412 [0.90 to 7.48] | 1.914 [0.72 to 3.91] | 1.679 [1.15 to 5.17]

20. Primary Outcome: Total Risperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the Secondary Peak
Description: Total risperidone concentration (risperidone and 9-hydroxyrisperidone) was determined by adding risperidone concentration to risperidone-equivalent concentration (obtained from the 9-hydroxyrisperidone data). Total risperidone concentration was calculated using the molecular weights of 410 for risperidone and 426 for 9-hydroxyrisperidone:
  * [Total Risperidone] = [Risperidone] + (410/426) * [9-hydroxyrisperidone]
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Secondary Peak, Injection 1 | 168.000 [23.83 to 504.00] | 264.000 [24.00 to 579.02] | 192.000 [24.00 to 574.30]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 228.000 [23.83 to 408.00] | 264.067 [24.00 to 408.00] | 216.000 [168.00 to 504.18]

21. Primary Outcome: Risperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24)
Description: AUC0-24 calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Initial Peak, Injection 1: number analyzed (Participants) | 14 | 15 | 15
  Initial Peak, Injection 1 | 103.8 [19.7 to 482.2] | 87.8 [30.0 to 367.9] | 99.5 [46.9 to 329.4]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 14 | 9
  Initial Peak, Injection 3 | 98.7 [35.1 to 557.9] | 107.1 [61.2 to 554.5] | 127.0 [82.1 to 329.2]

22. Primary Outcome: Risperidone PK: Maximum Plasma Concentration (Cmax) During Initial Peak
Description: Cmax determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Initial Peak, Injection 1 | 6.280 [1.32 to 25.70] | 5.460 [1.75 to 16.80] | 6.470 [2.80 to 15.30]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 4.955 [1.98 to 26.30] | 6.680 [2.89 to 30.60] | 7.145 [4.27 to 18.30]

23. Primary Outcome: Risperidone PK: Time of Maximum Plasma Concentration (Tmax) During Initial Peak
Description: Tmax determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Initial Peak, Injection 1 (Day 1 injection to 24 hours after injection)
  * Initial Peak, Injection 3 (Day 57 injection to 24 hours after injection)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Initial Peak, Injection 1 | 6.000 [3.00 to 23.83] | 6.000 [2.00 to 6.02] | 4.000 [1.00 to 6.00]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 6.000 [2.00 to 24.00] | 6.000 [3.00 to 24.08] | 4.483 [2.00 to 24.00]

24. Primary Outcome: Risperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to Time Tau (Where Tau=28 Days) (AUCtau)
Description: AUCtau calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 1250.9 [403.7 to 8706.0] | 1663.4 [764.3 to 10010.9] | 3099.4 [1768.5 to 7202.0]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 2144.6 [741.2 to 10490.3] | 2647.1 [1683.5 to 15384.8] | 3621.2 [2084.2 to 7812.0]

25. Primary Outcome: Risperidone PK: Average Plasma Concentration (Cavg) Over the PK Profile
Description: The average of plasma concentrations calculated as AUCtau/ tau (tau = 28 days)
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 1.861 [0.60 to 12.96] | 2.475 [1.14 to 14.90] | 4.612 [2.63 to 10.72]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 3.191 [1.10 to 15.61] | 3.939 [2.51 to 22.89] | 5.389 [3.10 to 11.62]

26. Primary Outcome: Risperidone PK: Maximum Plasma Concentration (Cmax) Over the PK Profile
Description: Maximum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 6.280 [1.32 to 37.40] | 7.520 [2.01 to 24.40] | 9.270 [4.27 to 18.50]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 5.720 [2.00 to 26.30] | 7.490 [4.23 to 38.40] | 12.125 [5.00 to 21.50]

27. Primary Outcome: Risperidone PK: Minimum Plasma Concentration (Cmin) Over the PK Profile
Description: Minimum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 0.829 [0.25 to 4.81] | 1.060 [0.42 to 9.44] | 1.720 [0.59 to 6.48]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 1.230 [0.39 to 4.24] | 2.100 [0.85 to 12.30] | 2.415 [1.24 to 4.83]

28. Primary Outcome: Risperidone PK: Percent Fluctuation Over the PK Profile
Description: The degree of fluctuation of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cavg, expressed as a percentage.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 190.745 [97.90 to 914.27] | 215.048 [100.42 to 423.52] | 173.609 [80.43 to 258.50]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 147.252 [75.60 to 212.01] | 140.688 [55.32 to 343.98] | 143.652 [93.11 to 206.70]

29. Primary Outcome: Risperidone PK: Swing Over the PK Profile
Description: The swing of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cmin.
  Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Overall, Injection 1 | 4.575 [1.58 to 34.19] | 4.151 [1.58 to 32.57] | 4.938 [1.33 to 12.06]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 4.077 [1.19 to 6.09] | 2.863 [0.77 to 10.56] | 3.159 [1.78 to 8.12]

30. Primary Outcome: Risperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the PK Profile
Description: Results are reported across two timeframes:
  * Overall, Injection 1 (Day 1 injection to Day 28)
  * Overall, Injection 3 (Day 57 injection to Day 84)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Overall, Injection 1 | 6.000 [4.00 to 408.28] | 168.000 [3.00 to 336.00] | 192.000 [3.00 to 384.95]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 18.000 [2.00 to 408.00] | 192.000 [3.00 to 671.75] | 180.000 [72.00 to 504.18]

31. Primary Outcome: Risperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Area Under the Plasma Concentration Curve (Rac(AUC))
Description: Accumulation index in terms of AUC calculated as ratio of AUCtau injection 3 / injection 1. Tau = 28 days.
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 14 | 10
ratio | 1.1 [0.6 to 4.8] | 1.7 [1.0 to 3.2] | 1.1 [1.0 to 1.9]

32. Primary Outcome: Risperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Maximum Plasma Concentrations (Rac(Cmax))
Description: Accumulation index in terms of Cmax calculated as ratio of Cmax injection 3 / injection 1.
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 15 | 10
ratio | 1.049 [0.20 to 2.16] | 1.214 [0.54 to 2.85] | 1.155 [0.62 to 1.59]

33. Primary Outcome: Risperidone PK: Area Under the Plasma Concentration-Time Curve From Day 2-29 Post Injection (AUC Day 2-29)
Description: Area under plasma concentration-time curve from 24 hours (Day 2) to the last quantifiable collection during dosing interval (28 days); calculated using the linear trapezoidal rule.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 15 | 13
  Secondary Peak, Injection 1 | 1198.2 [384.0 to 8450.7] | 1544.9 [730.6 to 9645.4] | 2937.3 [1133.1 to 6919.4]
  Secondary Peak, Injection 3: number analyzed (Participants) | 13 | 14 | 10
  Secondary Peak, Injection 3 | 2204.6 [836.0 to 9933.4] | 2494.8 [1621.8 to 14833.4] | 3476.6 [1996.8 to 7597.0]

34. Primary Outcome: Risperidone PK: Average Plasma Concentration Over the Secondary Peak (Cavg, Day 2-29)
Description: The average of plasma concentrations in the plateau, calculated as AUC Day 2-29/time
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 15 | 13
  Secondary Peak, Injection 1 | 1.849 [0.59 to 13.04] | 2.384 [1.13 to 14.88] | 4.533 [1.75 to 10.68]
  Secondary Peak, Injection 3: number analyzed (Participants) | 13 | 14 | 10
  Secondary Peak, Injection 3 | 3.402 [1.29 to 15.33] | 3.850 [2.50 to 22.89] | 5.365 [3.08 to 11.72]

35. Primary Outcome: Risperidone PK: Maximum Plasma Concentration Over the Secondary Peak (Cmax)
Description: Maximum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  Secondary Peak, Injection 1 (Day 2 - Day 29) Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 3.120 [0.76 to 37.40] | 5.950 [2.01 to 24.40] | 7.950 [2.98 to 18.50]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 5.220 [1.46 to 25.50] | 7.010 [4.23 to 38.40] | 12.125 [5.09 to 21.50]

36. Primary Outcome: Risperidone PK: Minimum Plasma Concentration (Cmin) Over the Secondary Peak
Description: Minimum plasma concentrations determined directly from individual concentration-time data.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 0.829 [0.25 to 4.81] | 1.070 [0.56 to 9.44] | 1.720 [0.59 to 6.48]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 1.230 [0.39 to 5.31] | 2.100 [0.85 to 12.30] | 2.415 [1.24 to 8.54]

37. Primary Outcome: Risperidone PK: Percent Fluctuation Over the Secondary Peak
Description: The degree of fluctuation of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cavg, expressed as a percentage.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 15 | 13
  Secondary Peak, Injection 1 | 134.805 [53.99 to 288.36] | 134.898 [68.79 to 274.33] | 141.030 [80.73 to 239.67]
  Secondary Peak, Injection 3: number analyzed (Participants) | 13 | 14 | 10
  Secondary Peak, Injection 3 | 136.691 [75.83 to 211.81] | 125.387 [55.36 to 345.51] | 138.380 [93.02 to 207.62]

38. Primary Outcome: Risperidone PK: Swing Over the Secondary Peak
Description: The swing of total risperidone plasma concentrations calculated as (Cmax - Cmin) / Cmin.
  Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Secondary Peak, Injection 1 | 2.644 [0.74 to 16.05] | 2.680 [0.94 to 8.52] | 3.813 [1.33 to 6.77]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 3.736 [1.09 to 6.09] | 2.652 [0.77 to 10.56] | 2.698 [1.52 to 8.12]

39. Primary Outcome: Risperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the Secondary Peak
Description: Results are reported across two timeframes:
  * Secondary Peak, Injection 1 (Day 2 - Day 29)
  * Secondary Peak, Injection 3 (Day 58 - Day 85)
  The PK sampling schedule was:
  * Days 1 and 57: within 15 minutes prior to dosing, and at 1, 2, 3, 4, 6, and 12 hours post-dose
  * Days 2, 4, 6, 8-12, 15, 18, 22, 25, 58, 60, 62, 64-68, 71, 74, 78, 81 once each day at same time of day as study drug administration
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Secondary Peak, Injection 1 | 120.000 [23.83 to 408.28] | 216.000 [24.02 to 336.00] | 192.000 [24.00 to 385.83]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 204.000 [23.83 to 576.00] | 216.00 [24.00 to 671.75] | 180.000 [72.00 to 504.18]

40. Primary Outcome: 9-hydroxyrisperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24)
Description: as for outcome 21
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Initial Peak, Injection 1: number analyzed (Participants) | 14 | 15 | 15
  Initial Peak, Injection 1 | 237.0 [149.4 to 407.6] | 251.1 [84.4 to 855.4] | 404.8 [152.4 to 715.0]
  Initial Peak, Injection 3: number analyzed (Participants) | 13 | 12 | 8
  Initial Peak, Injection 3 | 169.2 [76.6 to 291.0] | 263.4 [93.7 to 514.4] | 342.6 [231.4 to 477.0]

41. Primary Outcome: 9-hydroxyrisperidone PK: Maximum Plasma Concentration (Cmax) During Initial Peak
Description: as for outcome 22
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Initial Peak, Injection 1 | 11.100 [6.64 to 24.30] | 12.900 [4.17 to 37.80] | 17.500 [7.32 to 33.30]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 9.470 [4.64 to 15.10] | 12.900 [4.73 to 27.10] | 17.450 [10.60 to 27.40]

42. Primary Outcome: 9-hydroxyrisperidone PK: Time of Maximum Plasma Concentration (Tmax) During Initial Peak
Description: as for outcome 23
Time Frame: Day 1-2, Day 57-58
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Initial Peak, Injection 1 | 4.000 [0.00 to 24.00] | 6.000 [0.00 to 24.02] | 6.000 [0.00 to 24.00]
  Initial Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Initial Peak, Injection 3 | 24.000 [0.00 to 24.00] | 24.000 [23.83 to 24.08] | 24.000 [23.85 to 24.00]

43. Primary Outcome: 9-hydroxyrisperidone PK: Area Under the Plasma Concentration-Time Curve From Time Zero to Time Tau (Where Tau=28 Days) (AUCtau)
Description: as for outcome 24
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 4927.0 [2074.5 to 8428.4] | 5607.5 [1788.4 to 18485.5] | 9862.2 [6172.8 to 12526.6]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 5538.3 [2877.4 to 11191.6] | 8546.7 [3039.2 to 14534.1] | 11666.9 [8212.3 to 14354.6]

44. Primary Outcome: 9-hydroxyrisperidone PK: Average Plasma Concentration (Cavg) Over the PK Profile
Description: as for outcome 25
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 7.332 [3.09 to 12.54] | 8.344 [2.66 to 27.51] | 14.676 [9.19 to 18.64]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 8.242 [4.28 to 16.65] | 12.718 [4.52 to 21.63] | 17.361 [12.22 to 21.36]

45. Primary Outcome: 9-hydroxyrisperidone PK: Maximum Plasma Concentration (Cmax) Over the PK Profile
Description: as for outcome 26
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 12.300 [8.48 to 24.30] | 15.600 [4.17 to 39.20] | 22.400 [15.60 to 40.20]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 13.450 [6.34 to 32.40] | 21.200 [7.30 to 34.70] | 29.600 [19.40 to 37.80]

46. Primary Outcome: 9-hydroxyrisperidone PK: Minimum Plasma Concentration (Cmin) Over the PK Profile
Description: as for outcome 27
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Overall, Injection 1 | 3.940 [1.40 to 9.28] | 4.240 [2.14 to 19.10] | 6.690 [2.75 to 11.40]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 4.180 [1.29 to 8.11] | 6.580 [2.41 to 11.60] | 8.365 [3.60 to 12.50]

47. Primary Outcome: 9-hydroxyrisperidone PK: Percent Fluctuation Over the PK Profile
Description: as for outcome 28
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Overall, Injection 1: number analyzed (Participants) | 15 | 15 | 11
  Overall, Injection 1 | 120.024 [66.15 to 313.00] | 124.696 [73.07 to 193.81] | 142.828 [66.46 to 178.05]
  Overall, Injection 3: number analyzed (Participants) | 14 | 14 | 10
  Overall, Injection 3 | 121.077 [47.08 to 195.10] | 106.728 [80.34 to 174.90] | 122.701 [79.58 to 172.77]

48. Primary Outcome: 9-hydroxyrisperidone PK: Swing Over the PK Profile
Description: as for outcome 29
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Overall, Injection 1 | 1.984 [0.99 to 12.11] | 2.041 [0.89 to 5.72] | 2.633 [0.96 to 8.37]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 2.901 [0.63 to 8.24] | 2.142 [1.28 to 6.51] | 2.240 [1.36 to 7.97]

49. Primary Outcome: 9-hydroxyrisperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the PK Profile
Description: as for outcome 30
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Overall, Injection 1 | 168.000 [0.00 to 504.00] | 168.000 [0.00 to 579.02] | 192.000 [0.00 to 574.30]
  Overall, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Overall, Injection 3 | 216.000 [1.00 to 408.00] | 264.000 [24.00 to 336.00] | 216.000 [168.00 to 552.00]

50. Primary Outcome: 9-hydroxyrisperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Area Under the Plasma Concentration Curve (Rac(AUC))
Description: as for outcome 31
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 14 | 10
ratio | 1.1 [0.8 to 2.1] | 1.5 [1.0 to 2.8] | 1.2 [1.0 to 1.8]

51. Primary Outcome: 9-hydroxyrisperidone PK: Accumulation Index Between Injections 1 and 3 In Terms of Maximum Plasma Concentrations (Rac(Cmax))
Description: as for outcome 32
Time Frame: Day 1-28, Day 57-84
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 14 | 15 | 10
ratio | 0.997 [0.51 to 2.20] | 1.442 [0.74 to 2.51] | 1.076 [0.89 to 2.42]

52. Primary Outcome: 9-hydroxyrisperidone PK: Area Under the Plasma Concentration-Time Curve From Day 2-29 Post Injection (AUC Day 2-29)
Description: as for outcome 33
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hr*ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 4696.8 [1906.9 to 8095.4] | 5222.9 [1704.6 to 17634.8] | 7891.0 [5039.4 to 12116.0]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 9
  Secondary Peak, Injection 3 | 5388.2 [2775.2 to 10973.2] | 8311.7 [2943.9 to 14239.6] | 11786.5 [7982.8 to 13933.7]

53. Primary Outcome: 9-hydroxyrisperidone PK: Average Plasma Concentration Over the Secondary Peak (Cavg, Day 2-29)
Description: as for outcome 34
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 7.248 [2.94 to 12.49] | 8.060 [2.63 to 27.21] | 12.177 [7.78 to 18.70]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 9
  Secondary Peak, Injection 3 | 8.315 [4.28 to 16.93] | 12.827 [4.54 to 21.97] | 18.189 [12.32 to 21.50]

54. Primary Outcome: 9-hydroxyrisperidone PK: Maximum Plasma Concentration Over the Secondary Peak (Cmax)
Description: as for outcome 35
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 12.300 [6.15 to 21.50] | 15.600 [3.45 to 39.20] | 22.300 [15.60 to 40.20]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 13.450 [6.34 to 32.40] | 21.200 [7.30 to 34.70] | 29.600 [19.40 to 37.80]

55. Primary Outcome: 9-hydroxyrisperidone PK: Minimum Plasma Concentration (Cmin) Over the Secondary Peak
Description: as for outcome 36
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ng/mL
  Secondary Peak, Injection 1 | 3.940 [1.40 to 9.28] | 4.250 [2.14 to 19.10] | 7.060 [2.75 to 11.40]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 4.180 [1.45 to 8.11] | 7.660 [2.41 to 13.60] | 11.450 [6.76 to 12.00]

56. Primary Outcome: 9-hydroxyrisperidone PK: Percent Fluctuation Over the Secondary Peak
Description: as for outcome 37
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of average concentration
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
percentage of average concentration
  Secondary Peak, Injection 1: number analyzed (Participants) | 15 | 14 | 11
  Secondary Peak, Injection 1 | 112.945 [57.64 to 252.39] | 127.274 [47.14 to 183.19] | 141.300 [73.92 to 210.24]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 9
  Secondary Peak, Injection 3 | 106.055 [34.50 to 191.68] | 104.207 [58.02 to 139.50] | 101.956 [79.06 to 147.98]

57. Primary Outcome: 9-hydroxyrisperidone PK: Swing Over the Secondary Peak
Description: as for outcome 38
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: ratio
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
ratio
  Secondary Peak, Injection 1 | 1.936 [0.77 to 12.11] | 2.041 [0.56 to 4.54] | 2.633 [0.96 to 5.95]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 2.018 [0.46 to 8.24] | 1.991 [0.74 to 2.88] | 1.595 [1.12 to 4.31]

58. Primary Outcome: 9-hydroxyrisperidone PK: Time of the Maximum Plasma Concentration (Tmax) Over the Secondary Peak
Description: as for outcome 39
Time Frame: Day 2-29, Day 58-85
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
hours
  Secondary Peak, Injection 1 | 216.000 [24.00 to 504.00] | 168.000 [24.00 to 579.02] | 216.000 [24.00 to 574.30]
  Secondary Peak, Injection 3: number analyzed (Participants) | 14 | 15 | 10
  Secondary Peak, Injection 3 | 228.000 [24.00 to 408.00] | 264.000 [24.00 to 336.00] | 216.000 [168.00 to 552.00]

59. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Scores at Baseline and Days 28, 56, 84 and 106
Description: The switch from oral risperidone to RBP-7000 subcutaneous injections for efficacy markers used the PANSS scores. The PANSS assessment is a medical scale designed to measure symptom severity among patients with schizophrenia. Each item is rated on a scale of 1=absent to 7=extreme. PANSS consists of three components:
  * The General Psychopathology Scale consists of 16 questions with a total range of 16 (no schizophrenia symptoms) to 112 (extreme schizophrenia symptoms).
  * Both the Positive Scale and the Negative Scale consists of 7 questions with a total range of 7 (no schizophrenia symptoms) to 49 (extreme symptoms) on each scale.
  The PANSS range for assuring stability was a total PANSS General Psychopathology Scale score of 70 or less, with no score of 4 on any of the 7 questions in the Positive scale.
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline: General Psychopathology Scale | 27.0 [21 to 34] | 24.0 [21 to 32] | 27.0 [22 to 32]
  Baseline: Positive Scale | 13.0 [10 to 15] | 14.0 [8 to 17] | 13.0 [10 to 17]
  Baseline: Negative Scale | 15.0 [11 to 24] | 18.0 [9 to 23] | 18.0 [13 to 22]
  Day 28: General Psychopathology Scale: number analyzed (Participants) | 15 | 15 | 11
  Day 28: General Psychopathology Scale | 28.0 [19 to 33] | 26.0 [20 to 46] | 27.0 [22 to 40]
  Day 28: Positive Scale: number analyzed (Participants) | 15 | 15 | 11
  Day 28: Positive Scale | 13.0 [11 to 23] | 12.0 [8 to 24] | 12.0 [10 to 20]
  Day 28: Negative Scale: number analyzed (Participants) | 15 | 15 | 11
  Day 28: Negative Scale | 16.0 [11 to 22] | 17.0 [9 to 23] | 18.0 [12 to 22]
  Day 56: General Psychopathology Scale: number analyzed (Participants) | 15 | 15 | 10
  Day 56: General Psychopathology Scale | 28.0 [22 to 33] | 26.0 [20 to 34] | 25.0 [22 to 29]
  Day 56: Positive Scale: number analyzed (Participants) | 15 | 15 | 10
  Day 56: Positive Scale | 13.0 [9 to 22] | 13.0 [9 to 21] | 11.5 [10 to 14]
  Day 56: Negative Scale: number analyzed (Participants) | 15 | 15 | 10
  Day 56: Negative Scale | 17.0 [11 to 21] | 18.0 [8 to 25] | 17.5 [12 to 21]
  Day 84: General Psychopathology Scale: number analyzed (Participants) | 14 | 14 | 10
  Day 84: General Psychopathology Scale | 28.0 [20 to 34] | 25.0 [19 to 32] | 25.0 [22 to 29]
  Day 84: Positive Scale: number analyzed (Participants) | 14 | 14 | 10
  Day 84: Positive Scale | 13.5 [9 to 19] | 12.5 [8 to 18] | 12.5 [10 to 15]
  Day 84: Negative Scale: number analyzed (Participants) | 14 | 14 | 10
  Day 84: Negative Scale | 15.5 [11 to 21] | 17.5 [13 to 24] | 16.0 [12 to 24]
  Day 106: General Psychopathology Scale: number analyzed (Participants) | 15 | 14 | 14
  Day 106: General Psychopathology Scale | 26.0 [19 to 32] | 23.5 [19 to 34] | 26.5 [21 to 48]
  Day 106: Positive Scale: number analyzed (Participants) | 15 | 14 | 14
  Day 106: Positive Scale | 13.0 [10 to 18] | 12.0 [7 to 19] | 14.0 [10 to 28]
  Day 106: Negative Scale: number analyzed (Participants) | 15 | 14 | 14
  Day 106: Negative Scale | 14.0 [11 to 21] | 18.0 [13 to 23] | 18.0 [11 to 26]

60. Secondary Outcome: Clinical Global Impression (CGI) Scores (Severity of Illness and Global Improvement) at Baseline and Days 28, 56, 84 and 106
Description: The switch from oral risperidone to RBP-7000 subcutaneous injections for efficacy markers used CGI scores. The CGI is used in the assessment of global illness severity and change in clinical condition over time in psychiatric patients.
  Severity of illness is measured on a 7-point scale with 1=normal, not at all ill and 7=among the most extremely ill patients.
  Global improvement is measured on a 7-point scale with 1=very much improved, 4=no change and 7=very much worse as compared to the severity of illness at baseline.
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline: Severity of illness | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 3.00]
  Day 28: Severity of illness: number analyzed (Participants) | 15 | 15 | 11
  Day 28: Severity of illness | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 4.00] | 3.0 [3.00 to 4.00]
  Day 28: Global improvement: number analyzed (Participants) | 14 | 15 | 11
  Day 28: Global improvement | 4.0 [3.00 to 5.00] | 4.0 [3.00 to 6.00] | 4.0 [3.00 to 5.00]
  Day 56: Severity of illness: number analyzed (Participants) | 15 | 15 | 10
  Day 56: Severity of illness | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 4.00] | 3.0 [3.00 to 3.00]
  Day 56: Global improvement: number analyzed (Participants) | 15 | 15 | 10
  Day 56: Global improvement | 4.0 [4.00 to 5.00] | 4.0 [4.00 to 5.00] | 4.0 [4.00 to 4.00]
  Day 84: Severity of illness: number analyzed (Participants) | 14 | 14 | 10
  Day 84: Severity of illness | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 3.00]
  Day 84: Global improvement: number analyzed (Participants) | 14 | 14 | 10
  Day 84: Global improvement | 4.0 [3.00 to 4.00] | 4.0 [3.00 to 5.00] | 4.0 [4.00 to 4.00]
  Day 106: Severity of illness: number analyzed (Participants) | 15 | 14 | 14
  Day 106: Severity of illness | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 3.00] | 3.0 [3.00 to 5.00]
  Day 106: Global improvement: number analyzed (Participants) | 15 | 14 | 14
  Day 106: Global improvement | 4.0 [2.00 to 4.00] | 4.0 [3.00 to 5.00] | 4.0 [3.00 to 6.00]

61. Secondary Outcome: Global Assessment of the Abnormal Involuntary Movement Scale (AIMS) for Tardive Dyskinesia at Baseline and Days 28, 56, 84 and 106
Description: The switch from oral risperidone to RBP-7000 subcutaneous injections for safety markers used AIMS. The AIMS is a scale that aids in the early detection and ongoing monitoring of tardive dyskinesia, a movement disorder that can result from long-term treatment with antipsychotic medication. By assessing the participant's body movement in specific positions requiring rotation, a psychiatrist is able to determine whether abnormal facial or body movements exist.
  The total score is the sum of 7 questions assessing movement plus 3 questions representing global assessments on the overall level of involuntary movement severity, incapacitation due to involuntary movement, and patient's awareness of involuntary movement. Each of the 10 questions are scored on a 0 (none) - 4 (extremely severe) scale. Plus two dental status questions are scored on a 0 (no) - 1 (yes) scale. The total score is therefore a scale of 0 (normal) - 42 (advanced tardive dyskinesia).
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 1.0 [0 to 12] | 0.0 [0 to 2] | 1.0 [0 to 5]
  Day 28: number analyzed (Participants) | 15 | 15 | 11
  Day 28 | 1.0 [0 to 12] | 0.0 [0 to 4] | 1.0 [0 to 6]
  Day 56: number analyzed (Participants) | 15 | 15 | 10
  Day 56 | 1.0 [0 to 12] | 0.0 [0 to 2] | 1.0 [0 to 6]
  Day 84: number analyzed (Participants) | 14 | 14 | 10
  Day 84 | 0.5 [0 to 12] | 0.0 [0 to 4] | 1.0 [0 to 5]
  Day 106: number analyzed (Participants) | 15 | 14 | 14
  Day 106 | 1.0 [0 to 12] | 0.0 [0 to 5] | 0.5 [0 to 5]

62. Secondary Outcome: Total Simpson-Angus Scale (SAS) Score at Baseline and Days 28, 56, 84 and 106
Description: The switch from oral risperidone to RBP-7000 subcutaneous injections for safety markers used SAS. The SAS is a 10-item scale used to detect the presence of drug induced parkinsonism and extrapyramidal side effects, and evaluates symptom severity. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0 to 4 scale with 0=normal and 4=extreme description of the particular side effect. The total range is 0=no side effects observed to 40 = extreme of each of the 10 side effects.
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 2]
  Day 28: number analyzed (Participants) | 15 | 15 | 11
  Day 28 | 0.0 [0 to 0] | 0.0 [0 to 3] | 0.0 [0 to 1]
  Day 56: number analyzed (Participants) | 15 | 15 | 10
  Day 56 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 1]
  Day 84: number analyzed (Participants) | 14 | 14 | 10
  Day 84 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 1]
  Day 106: number analyzed (Participants) | 15 | 14 | 14
  Day 106 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 1]

63. Secondary Outcome: Global Clinical Assessment of Akathisia Using the Barnes Akathisia Scale (BAS) at Baseline and Days 28, 56, 84 and 106
Description: The BAS is a scale that detects the presence and severity of any drug induced akathisia. The scale measures objective and subjective effects such as restlessness and awareness of restlessness, respectively. Participants are observed while seated, then while standing and engaged in neutral conversation. Symptoms observed during additional situations, such as participant behavior on the ward, may also be rated. Subjective phenomena should be elicited through direct questioning of the participant. The global clinical assessment is reported on a scale of 0 to 5, where 0 = absent and 5 = severe akathisia.
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 1]
  Day 28: number analyzed (Participants) | 15 | 15 | 11
  Day 28 | 0.0 [0 to 2] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 56: number analyzed (Participants) | 15 | 15 | 10
  Day 56 | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Day 84: number analyzed (Participants) | 14 | 14 | 10
  Day 84 | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Day 106: number analyzed (Participants) | 15 | 14 | 14
  Day 106 | 0.0 [0 to 2] | 0.0 [0 to 0] | 0.0 [0 to 1]

64. Secondary Outcome: Participants With Suicidal Ideation or Behavior as Identified Using the Columbia-Suicide Severity Rating Scale (C-SSRS) Score at Baseline and Days 28, 56, 84 and 106
Description: The C-SSRS is a scale developed by the National Institute of Mental Health trial group as a counterpart to the FDA's categorization of suicidal events. It was developed by a careful review and consequent categorization of thoughts and behavior that were statistically identified as significantly related to suicidal behavior. The scale captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors throughout lifetime at screening, baseline, and for the time interval since last administration for repeat administrations during a study.
  This outcome reports the number of participants with suicidal ideation or behavior.
Time Frame: Baseline (Day -1), Days 28, 56, 84, and End of Study (Day 106 or early termination visit)
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Baseline: Suicidal ideation or behavior | 0 | 0 | 0
  Day 28: Suicidal ideation or behavior: number analyzed (Participants) | 15 | 15 | 11
  Day 28: Suicidal ideation or behavior | 0 | 1 | 1
  Day 56: Suicidal ideation or behavior: number analyzed (Participants) | 15 | 15 | 10
  Day 56: Suicidal ideation or behavior | 1 | 0 | 0
  Day 84: Suicidal ideation or behavior: number analyzed (Participants) | 14 | 14 | 10
  Day 84: Suicidal ideation or behavior | 0 | 0 | 0
  Day 106: Suicidal ideation or behavior: number analyzed (Participants) | 15 | 14 | 14
  Day 106: Suicidal ideation or behavior | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 106
Arm/Group | Cohort 1, RBP-7000 60 mg | Cohort 2, RBP-7000 90 mg | Cohort 3, RBP-7000 120 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 11/15 | 11/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, RBP-7000 60 mg (N=15) | Cohort 2, RBP-7000 90 mg (N=15) | Cohort 3, RBP-7000 120 mg (N=15)
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, RBP-7000 60 mg (N=15) | Cohort 2, RBP-7000 90 mg (N=15) | Cohort 3, RBP-7000 120 mg (N=15)
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Influenza-like illness (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight increased (Investigations) | 4 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 3 | 1
Extrapyramidal disorder (Nervous system disorders) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1
Drooling (Nervous system disorders) | 1 | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Dermititis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multicenter publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.